CLINICAL TRIAL: NCT01355081
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase III Study to Assess the Efficacy and Safety of Lu AA21004 in Patients With Major Depressive Disorder
Brief Title: Efficacy Study of Vortioxetine (Lu AA21004) for Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LuAA21004/CCT-003; U1111-1120-9277 (Registry Identifier: WHO); JapicCTI-111492 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Results first posted 2014-11-11 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Major Depressive Disorder
Keywords: Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vortioxetine 5 mg (Experimental): Vortioxetine 5 mg, tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Vortioxetine
- Vortioxetine 10 mg (Experimental): Vortioxetine 10 mg, tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Vortioxetine
- Placebo (Placebo Comparator): Vortioxetine placebo-matching tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine tablets
  Other Names: Lu AA21004; BRINTELLIX
  Arms: Vortioxetine 10 mg; Vortioxetine 5 mg
Drug: Placebo — Vortioxetine placebo
  Other Names: Vortioxetine placebo-matching tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of 8-week treatment with Vortioxetine (Lu AA21004), once daily (QD), in Japanese participants with major depressive disorder.

The purpose of this study is to assess the efficacy, safety and tolerability of 8-week treatment with Lu AA21004, once daily (QD), in Japanese participants with major depressive disorder.

DETAILED DESCRIPTION:
Lu AA21004 was discovered by H. Lundbeck A/S, and is under co-development by H. Lundbeck A/S and Takeda for the treatment of major depressive disorder and general anxiety disorder. Major depressive disorder (MDD) is a chronic, recurring disease with considerable morbidity in the general population. The estimated lifetime prevalence of major depression in the adult population is 5 to 25%, with approximately 2-fold higher prevalence in women than in men. The hallmark of the disease is a depressed mood, with additional symptoms including sleep disturbances, psychomotor agitation or retardation, sexual dysfunction, weight loss, concentration difficulties and delusional ideas. In addition to direct ill effects, MDD causes suicide or job loss and exerts indirect influence on social economy. This study will assess the efficacy and the safety of Lu AA21004. This study consists of a 1-week screening period, an 8-week double-blind treatment period, 4-week safety follow-up.The duration of the study is 13 weeks in total. Blood samples will be collected from participants, and a safety follow-up contact (visit or phone call) will be made 4 weeks after completion of the 8-week double-blind treatment period. Subjects who complete the 8-week double-blind treatment period can successively enter a long-term extension study (Lu AA21004/OCT-001; NCT01395147; hereinafter, OCT-001), if they meet all inclusion criteria and none of exclusion criteria of the OCT-001 study and are willing to participate in the OCT-001 study. Subjects who will enter the OCT-001 will not be requested to safety follow-up after completion of the 8-week double-blind treatment period.

Lu AA21004 was discovered by H. Lundbeck A/S, and is under co-development by H. Lundbeck A/S and Takeda for the treatment of major depressive disorder and general anxiety disorder.

Major depressive disorder (MDD) is a chronic, recurring disease with considerable morbidity in the general population. The estimated lifetime prevalence of major depression in the adult population is 5 to 25%, with approximately 2-fold higher prevalence in women than in men. The hallmark of the disease is a depressed mood, with additional symptoms including sleep disturbances, psychomotor agitation or retardation, sexual dysfunction, weight loss, concentration difficulties and delusional ideas. In addition to direct ill effects, MDD causes suicide or job loss and exerts indirect influence on social economy.

This study will assess the efficacy and the safety of Lu AA21004. This study consists of a 1-week screening period, an 8-week double-blind treatment period, 4-week s safety follow-up.The duration of the study is 13 weeks in total. Blood samples will be collected from participants, and a safety follow-up contact (visit or phone call) will be made 4 weeks after completion of the 8-week double-blind treatment period.

Subjects who complete the 8-week double-blind treatment period can successively enter a long-term extension study (Lu AA21004/OCT-001; NCT01395147; hereinafter, OCT-001), if they meet all inclusion criteria and none of exclusion criteria of the OCT-001 study and are willing to participate in the OCT-001 study.

Subjects who will enter the OCT-001 will not be requested to safety follow-up after completion of the 8-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. The subject suffers from Major Depressive Disorder (MDD) as the primary diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria (classification code 296.2x and 296.3x).
2. The reported duration of the current major depressive episode is at least 3 months at the Screening Visit.
3. The subject has a Montgomery-Åsberg Depression Rating Scale (MADRS) total score ≥26 at the Screening and Baseline Visits.
4. The subject has a Clinical Global Impression Scale-Severity (CGI-S) score ≥4 at the Screening and Baseline Visits

Exclusion Criteria:

1. The subject has one or more of the following conditions:

   * Any current psychiatric disorder other than MDD as defined in the DSM-IV-TR. A subject who exhibits symptoms of anxiety is eligible unless the subject fulfills the diagnostic criteria for a current anxiety disorder per DSM-IV-TR.
   * Current diagnosis or history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
   * Current diagnosis or history of any substance-related disorder (except nicotine and caffeine-related disorders) as defined in the DSM-IV-TR.
   * Presence or history of a clinically significant neurological disorder (including epilepsy).
   * Neurodegenerative disorder (Alzheimer's disease, Parkinson's disease, multiple sclerosis, Huntington's disease, etc.).
   * Any DSM-IV-TR axis II disorder that might compromise the study.
2. The current depressive symptoms of the subject are considered by the investigator to have been resistant to 2 adequate antidepressant treatments of at least 6 weeks duration each.
3. The subject is at significant risk of suicide or has a score ≥5 on Item 10 (suicidal thoughts) of the MADRS at the Screening and Baseline Visit, or has attempted suicide within 6 months prior to the Screening Visit.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Manager, Study Director — Takeda
Locations (32):
- Japan (32):
  - Inzai-shi, Chiba
  - Noda, Chiba
  - Fukuoka, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Annaka-shi, Gunma
  - Fujioka-shi, Gunma
  - Takasaki-shi, Gunma
  - Hatsukaichi-shi, Hiroshima
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Amagasaki-shi, Hyōgo
  - Kobe, Hyōgo
  - Ibaraki, Ibaraki
  - Fujisawa-shi, Kanagawa
  - Kawasaki-shi, Kanagawa
  - Sagamihara-shi, Kanagawa
  - Yokohama, Kanagawa
  - Osaka, Kita-ku
  - Kumamoto, Kumamoto
  - Kyoto, Kyoto
  - Kurashiki-shi, Okayama-ken
  - Osaka, Osaka
  - Fukaya-shi, Saitama
  - Saitama, Saitama
  - Utsunomiya, Tochigi
  - Anan-shi, Tokushima
  - Tokushisma-shi, Tokushima
  - Hachioji-shi, Tokyo
  - Katsushika-ku, Tokyo
  - Musashino-shi, Tokyo
  - Tokyo, Tokyo
  - Nanyo-shi, Yamagata

REFERENCES:
- [Derived] Inoue T, Nishimura A, Sasai K, Kitagawa T. Randomized, 8-week, double-blind, placebo-controlled trial of vortioxetine in Japanese adults with major depressive disorder, followed by a 52-week open-label extension trial. Psychiatry Clin Neurosci. 2018 Feb;72(2):103-115. doi: 10.1111/pcn.12623. Epub 2017 Dec 27. PMID 29160598

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 32 investigative sites throughout Japan from 13 May 2011 to 21 December 2012.
Pre-assignment Details: Participants with a diagnosis of major depressive disorder were enrolled equally in 1 of 3 treatment groups: once a day 5 mg or 10 mg vortioxetine (Lu AA21004) or placebo.
Period: Overall Study
Arm/Group | Vortioxetine 5 mg | Vortioxetine 10 mg | Placebo
Started | 119 | 123 | 124
Completed | 112 | 113 | 113
Not Completed | 7 | 10 | 11
Not completed — Pretreatment Event or Adverse Event | 3 | 4 | 6
Not completed — Major Protocol Deviation | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal of Consent | 2 | 3 | 3
Not completed — Lack of Efficacy | 2 | 1 | 1
Not completed — Non Compliance with Study Medication | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vortioxetine 5 mg | Vortioxetine 10 mg | Placebo | Total
Number analyzed (Participants) | 119 | 123 | 124 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (10.85) | 38.8 (10.99) | 37.6 (10.67) | 38.4 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 54 | 67 | 171
  Male | 69 | 69 | 57 | 195
Region of Enrollment [Number; unit: participants]
  Japan | 119 | 123 | 124 | 366
Height [Mean (Standard Deviation); unit: cm] | 165.7 (8.45) | 165.6 (8.51) | 163.9 (8.46) | 165.1 (8.49)
Weight [Mean (Standard Deviation); unit: kg] | 62.18 (11.357) | 62.11 (15.883) | 60.86 (12.690) | 61.71 (13.441)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.59 (3.366) | 22.42 (4.306) | 22.57 (4.016) | 22.53 (3.911)
Cytochrome p450 (CYP)2D6 Phenotype [Number; unit: participants]
  Ultra-rapid Metabolizer (UM) | 1 | 1 | 2 | 4
  Extensive Metabolizer (EM) | 91 | 97 | 96 | 284
  Intermediate Metabolizer (IM) | 25 | 20 | 21 | 66
  Poor Metabolizer (PM) | 0 | 1 | 0 | 1
  Unknown | 2 | 4 | 5 | 11
Smoking Classification [Number; unit: participants]
  Current smoker | 39 | 41 | 40 | 120
  Ex-smoker | 26 | 24 | 24 | 74
  Never Smoked | 54 | 58 | 60 | 172
History of Alcohol Consumption [Number; unit: participants]
  Never | 34 | 32 | 41 | 107
  Once Monthly or Less Often | 33 | 40 | 40 | 113
  Once a Week | 16 | 20 | 20 | 56
  2 to 6 Times/Week | 21 | 20 | 15 | 56
  Daily | 15 | 11 | 8 | 34
Status of Major Depressive Episode (MDE) [Number; unit: participants] — An MDE is a period marked by depressed mood, loss of interest or pleasure, disturbed sleep or appetite, low energy, feelings of guilt or low self-worth, and poor concentration.
  participants
    Single episode | 70 | 68 | 76 | 214
    Recurrent episode | 49 | 55 | 48 | 152
Pharmacotherapy for Current Major Depressive Episode [Number; unit: participants]
  Yes | 68 | 68 | 74 | 210
  No | 51 | 55 | 50 | 156
Montgomery Åsberg Depression Rating Scale (MADRS) Total Score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  scores on a scale | 32.2 (4.81) | 32.5 (4.93) | 32.5 (4.50) | 32.4 (4.74)
Hamilton Depression Scale (HAM-D17) Total Score [Mean (Standard Deviation); unit: scores on a scale] — The HAM-D17 is a clinician-rated scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 52 where a higher score indicates a greater depressive state.
  scores on a scale | 20.9 (4.12) | 21.2 (4.43) | 21.5 (4.48) | 21.2 (4.34)
Clinical Global Impression - Severity Scale Score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  scores on a scale | 4.5 (0.65) | 4.5 (0.64) | 4.6 (0.69) | 4.5 (0.66)
Sheehan Disability Scale (SDS) - Total Score [Mean (Standard Deviation); unit: scores on a scale] — The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment.
  scores on a scale | 15.5 (6.12) | 15.2 (5.97) | 15.4 (5.45) | 15.4 (5.83)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score After 8 Weeks of Treatment
Description: MADRS is a 10-item clinician rated scale that measures overall severity of depressive symptoms (such as apparent sadness, reported sadness, inner tension) rated on a 7-point Likert scale from 0 (symptoms absent) to 6 (severe depression) with a total possible score range from 0 to 60. Higher scores indicate greater severity of symptoms. A negative change from Baseline indicates that symptoms have improved. An analysis of covariance (ANCOVA) model was used with change in MADRS total score as a dependent variable, treatment as a fixed effect and the baseline MADRS total score as a covariate.
Time Frame: Baseline, Week 8
Population: Participants from the Full Analysis Set (FAS), defined as all participants who were randomized and received at least 1 dose of study drug; who had data available for this outcome measure. One participant in the Vortioxetine 10 mg group was excluded due to a major protocol deviation. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vortioxetine 5 mg | Vortioxetine 10 mg | Placebo
Number analyzed (Participants) | 119 | 122 | 123
scores on a scale | -15.84 (0.885) | -14.85 (0.874) | -13.81 (0.870)
Statistical Analysis 1: Comparison: Vortioxetine 5 mg vs Placebo; Test type: Superiority or Other; p = 0.1031, ANCOVA; Change in MADRS total score as a dependent variable, treatment as a fixed effect and the baseline MADRS total score as a covariate; Least square means difference = -2.03, 95% CI 2-sided [-4.467 to 0.413], Standard Error of Mean 1.241
Statistical Analysis 2: Comparison: Vortioxetine 10 mg vs Placebo; Test type: Superiority or Other; p = 0.4008, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least square mean difference = -1.04, 95% CI 2-sided [-3.461 to 1.387], Standard Error of Mean 1.233

2. Secondary Outcome: Percentage of Patients With MADRS Response After 8 Weeks of Treatment
Description: MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (such as apparent sadness, reported sadness, inner tension) rated on a 7-point Likert scale from 0 (symptoms absent) to 6 (severe depression) with a total possible score range from 0 to 60. Higher scores indicate greater severity of symptoms. Response is defined as a ≥50% decrease in the MADRS Total Score from Baseline.
Time Frame: Baseline, Week 8
Population: Participants from the Full Analysis Set (FAS), defined as all participants who were randomized and received at least 1 dose of study drug, who had data available for this outcome measure. One participant in the Vortioxetine 10 mg group was excluded due to a major protocol deviation.
Measure: Number; unit: percentage of participants
Arm/Group | Vortioxetine 5 mg | Vortioxetine 10 mg | Placebo
Number analyzed (Participants) | 119 | 122 | 123
percentage of participants | 51.3 | 45.9 | 39.8

3. Secondary Outcome: Percentage of Patients With MADRS Remission After 8 Weeks of Treatment
Description: MADRS is a 10-item clinician rated scale to measure overall severity of depressive symptoms (such as apparent sadness, reported sadness, inner tension) rated on a 7-point Likert scale from 0 (symptoms absent) to 6 (severe depression) with a total possible score range from 0 to 60. Higher scores indicate greater severity of symptoms. Remission is defined as a MADRS Total Score ≤10.
Time Frame: Week 8
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Vortioxetine 5 mg | Vortioxetine 10 mg | Placebo
Number analyzed (Participants) | 119 | 122 | 123
percentage of participants | 29.4 | 28.7 | 22.0

4. Secondary Outcome: Change From Baseline in the Hamilton Depression Scale (HAM-D17) Total Score After 8 Weeks of Treatment
Description: The HAM-D17 is a 17-item rating scale that assesses depressed mood, agitation and somatic symptoms of depression, rated on a 5-point scale from 0 (absent) to 4 (very severe) with a total score range from 0 to 52. Higher scores indicate greater severity of depression symptoms. A negative change from Baseline indicates that symptoms have improved. ANCOVA model was used with treatment as a fixed effect and the baseline HAM-D17 score as a covariate.
Time Frame: Baseline, Week 8
Population: Participants from the Full Analysis Set (FAS), defined as all participants who were randomized and received at least 1 dose of study drug, who had data available for this outcome measure. One participant in the Vortioxetine 10 mg group was excluded due to a major protocol deviation. Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vortioxetine 5 mg | Vortioxetine 10 mg | Placebo
Number analyzed (Participants) | 119 | 121 | 122
scores on a scale | -9.56 (0.586) | -8.54 (0.580) | -8.40 (0.578)

5. Secondary Outcome: Clinical Global Impression Scale-Improvement (CGI-I) Score After 8 Weeks of Treatment
Description: The CGI-I assesses the clinician's impression of the participant's state of mental illness improvement and consists of one question for the investigator: "Compared to his condition at the start of the study, how much has this patient changed?" which is rated on a seven-point scale (1=very much improved; 2=much improved; 3=minimally improved; 4=no change from baseline; 5=minimally worse; 6= much worse; 7=very much worse). Higher scores indicate greater severity of illness. Values closest to 1 for this outcome measure indicate the greatest improvement of symptoms. ANCOVA model was used with treatment as a fixed effect and the baseline CGI-Severity (CGI-S) score as a covariate.
Time Frame: Baseline, Week 8
Population: Participants from the Full Analysis Set (FAS), defined as all participants who were randomized and received at least 1 dose of study drug, who had data available for this outcome measure. One participant in the Vortioxetine 10 mg group was excluded due to a major protocol deviation. Last Observation Carried Forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vortioxetine 5 mg | Vortioxetine 10 mg | Placebo
Number analyzed (Participants) | 119 | 122 | 123
scores on a scale | 2.44 (0.100) | 2.57 (0.099) | 2.66 (0.099)

6. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score After 8 Weeks of Treatment
Description: The SDS is a 3 item rating scale to assess functional impairment (panic, anxiety, phobic and depressive symptoms) over three inter-related domains (work/school, social life, and family life/home responsibilities) rated on an 11 point scale from 0 (not at all) to 10 (extremely) with a total score range from 0 to 30. Higher scores indicate greater severity of impairment. A negative change from Baseline indicates that symptoms have improved. ANCOVA model was used with treatment as a fixed effect and the Baseline SDS total score as a covariate.
Time Frame: Baseline, Week 8
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vortioxetine 5 mg | Vortioxetine 10 mg | Placebo
Number analyzed (Participants) | 119 | 121 | 122
scores on a scale | -5.01 (0.510) | -4.02 (0.506) | -2.91 (0.504)

ADVERSE EVENTS:
Time Frame: 8-week double blind treatment period and 4-week follow-up safety period, or up to 4 weeks after withdrawal visit, excluding those who enrolled in the long-term extension study (Up to 12 Weeks)
Description: At each visit the investigator documented adverse events and abnormal laboratory findings reported by the patient or observed by the investigator irrespective of relation to study drug. Safety analysis set included all participants who received study drug. 1 participant in the Vortioxetine 10 mg group was excluded due to a major protocol violation.
Arm/Group | Vortioxetine 5 mg | Vortioxetine 10 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/119 | 1/122 | 1/124
Other Adverse Events (participants affected / at risk) | 80/119 | 93/122 | 78/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine 5 mg (N=119) | Vortioxetine 10 mg (N=122) | Placebo (N=124)
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine 5 mg (N=119) | Vortioxetine 10 mg (N=122) | Placebo (N=124)
Nausea (Gastrointestinal disorders) | 20 | 35 | 9
Diarrhoea (Gastrointestinal disorders) | 10 | 13 | 10
Nasopharyngitis (Infections and infestations) | 24 | 17 | 21
Somnolence (Nervous system disorders) | 7 | 12 | 9
Headache (Nervous system disorders) | 10 | 6 | 8
Suicidal ideation (Psychiatric disorders) | 1 | 8 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 0
Motion sickness (Ear and labyrinth disorders) | 0 | 1 | 0
Asthenopia (Eye disorders) | 0 | 1 | 0
Blepharospasm (Eye disorders) | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1
Ocular hypertension (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 5 | 4
Vomiting (Gastrointestinal disorders) | 3 | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0 | 1
Toothache (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0
Thirst (General disorders) | 3 | 5 | 3
Feeling abnormal (General disorders) | 0 | 2 | 2
Fatigue (General disorders) | 0 | 3 | 0
Malaise (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Facial pain (General disorders) | 0 | 1 | 0
Irritability (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 3
Gastroenteritis (Infections and infestations) | 0 | 0 | 3
Oral herpes (Infections and infestations) | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0
Otitis media chronic (Infections and infestations) | 1 | 0 | 0
Pericoronitis (Infections and infestations) | 0 | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 1 | 0
Viral rash (Infections and infestations) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 5 | 1 | 5
Blood triglycerides increased (Investigations) | 3 | 0 | 5
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1
Liver function test abnormal (Investigations) | 1 | 2 | 1
Blood bilirubin increased (Investigations) | 1 | 2 | 0
Blood uric acid increased (Investigations) | 1 | 1 | 0
Blood urine present (Investigations) | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 0
Glucose urine present (Investigations) | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 5 | 2
Dizziness postural (Nervous system disorders) | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 1
Nightmare (Psychiatric disorders) | 0 | 2 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0 | 0
Self injurious behaviour (Psychiatric disorders) | 1 | 0 | 0
Suicidal behaviour (Psychiatric disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Menstruation irregular (Reproductive system and breast disorders) | 1 | 0 | 0
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.